CLINICAL TRIAL: NCT07279207
Title: Prospective Analysis of Cardiac Electrostimulation and Atrial Fibrillation (PACE-AF)
Brief Title: PACE-AF: Prospective Analysis of Cardiac Electrostimulation and Atrial Fibrillation
Acronym: PACE-AF
Status: Not yet recruiting | Type: Observational
Sponsor: Ilya Lukin (Other)
Responsible Party: Sponsor
Other Study IDs: PACE-AF
Record Dates: First submitted 2025-11-19; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation; Sick Sinus Syndrome; Atrioventricular Block
Keywords: Pacemaker; Dual-chamber pacing; Pacemaker algorithms; Conduction system pacing; His bundle pacing; Left bundle branch pacing; Catheter ablation; Cryoablation; Arrhythmia prevention
MeSH Terms: conditions — Atrial Fibrillation; Sick Sinus Syndrome; Atrioventricular Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PACE-AF is a prospective, observational patient registry designed to evaluate the impact of pacemaker algorithms on atrial fibrillation (AF) incidence, progression, and clinical outcomes in patients implanted with dual-chamber pacemakers. The registry aims to include 400-500 patients with longitudinal follow-up. Primary outcomes are progression to permanent AF and all-cause mortality. Secondary outcomes include quality of life, hospitalization, and cardiovascular events.

DETAILED DESCRIPTION:
The PACE-AF registry is a prospective, observational study designed to systematically evaluate the influence of advanced pacemaker algorithms on atrial fibrillation (AF) development and progression. Algorithms of interest include atrial preventive pacing, atrial tachycardia termination, Antitachycardia Pacing (reactive ATP), and other vendor-specific features. The registry will consecutively enroll all patients receiving dual-chamber pacemakers at Tver State Medical University and associated clinical sites.

Approximately 400-500 patients are planned for inclusion, with follow-up scheduled according to standard of care and device interrogation. Primary outcomes are progression to permanent AF and all-cause mortality. Secondary outcomes include hospitalization, cardiovascular events, and quality of life.

In addition, predefined substudies will investigate the hemodynamic consequences of different pacing sites (apical right ventricular pacing, septal pacing, His bundle pacing, and left bundle branch pacing). Hemodynamic evaluation will be performed intraoperatively using echocardiography, invasive atrial pressure monitoring, and electroanatomical mapping techniques. Further exploratory analyses will assess outcomes in pacemaker patients who have undergone catheter ablation or cryoablation for AF.

This registry represents a structured attempt to combine real-world data on pacemaker function with detailed hemodynamic and electrophysiological assessment, with the overarching aim of identifying strategies to prevent AF progression in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years

  * Implantation of a dual-chamber permanent pacemaker
  * Ability to provide informed consent
  * Willingness to participate in long-term follow-up

Exclusion Criteria:

* • Single-chamber pacemaker or Cardiac Resynchronization Therapy device at baseline

  * Life expectancy < 1 year due to non-cardiac comorbidities
  * Inability to comply with follow-up visits or device interrogation
  * Participation in another clinical trial that could interfere with study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients undergoing implantation of dual-chamber pacemakers at Tver State Medical University and affiliated hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Permanent Atrial Fibrillation (%) | Up to 3 years of follow-up
  Transition from paroxysmal or persistent atrial fibrillation to permanent atrial fibrillation, defined as a clinical decision to cease rhythm control strategies and accept permanent AF

SECONDARY OUTCOMES:
All-Cause Mortality Rate (number of participants) | Up to 3 years
  Death from any cause during follow-up, according to clinical documentation and death registry data
AF Burden (% of time in atrial fibrillation) | Up to 3 years
  Percentage of time in atrial fibrillation recorded by device diagnostics (atrial high-rate episodes / AT/AF detection)
Mean Left Atrial Pressure During Pacing (mmHg) | Baseline intraoperative
  Intraoperative measurement of mean left atrial pressure according to pacing site.
Change in Left Atrial Volume Index (mL/m²) | Baseline intraoperative + up to 12 months follow-up
  Change from baseline in left atrial volume index measured by transthoracic echocardiography according to pacing site.

CONTACTS AND LOCATIONS:
Overall Officials: Ilya B. Lukin, MD, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Tver State Medical University Clinical Center, Tver', Tver Oblast, Russia

IPD SHARING:
Plan to Share IPD: No
No, but available on request

REFERENCES:
- [Background] Lukin I.B., Federiakin D.V., Gridiakina D.I., Karaagach M.H. The effect of atrial pacing on the risk of atrial tachyarrhythmias in patients with dual-chamber cardiac pacemakers: a pilot study. Journal of Arrhythmology. 2025;32(3):45-50. (In Russ.) https://doi.org/10.35336/VA-1509
- See also: Author Open Researcher and Contributor ID (ORCID Profile) (Ilya B. Lukin) — http://orcid.org/0000-0003-1871-2754
- See also: Pilot study on atrial pacing algorithms and atrial fibrillation (Lukin et al., 2025) — http://doi.org/10.35336/VA-1509